CLINICAL TRIAL: NCT00496080
Title: A Pivotal Study of Doppler Guided Uterine Artery Occlusion as Treatment for the Reduction of Fibroid Associated Bleeding
Brief Title: Doppler-Guided Uterine Artery Occlusion (DUAO) Device for Fibroid Related Bleeding
Acronym: DUAO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial terminated early due to results from a similar study.
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300-06-004
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2012-07-24 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Menorrhagia; Uterine Fibroids
Keywords: Menorrhagia associated with Uterine Fibroids
MeSH Terms: conditions — Menorrhagia; Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DUAO Device (Experimental): Doppler-guided uterine artery occlusion device (Single-arm study)
  Interventions: Device: Doppler-Guided Uterine Artery Occlusion Device (DUAO)

INTERVENTIONS:
Device: Doppler-Guided Uterine Artery Occlusion Device (DUAO) — Investigational transvaginal clamp inserted one time for 6 hours.
  Other Names: floSTAT

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of Doppler guided uterine artery occlusion (D-UAO) for the reduction of fibroid associated bleeding.

DETAILED DESCRIPTION:
The GYNECARE GYNOCCLUDE D-UAO Instruments are single-use disposable instruments consisting of a GYNECARE GYNOCCLUDE Uterine Stabilizer, a GYNECARE GYNOCCLUDEM Introducer Sheath, a GYNECARE GYNOCCLUDE Doppler Clamp, and a GYNECARE GYNOCCLUDE Coupler.

ELIGIBILITY:
Inclusion Criteria:

* 25 to 50 years of age;
* PBLAC score of 150 or greater;
* Completed child-bearing;
* Normal Pap smear within 12 months;
* Cervix suitable for tenaculum placement as determined by pelvic exam;
* At least one uterine fibroid of 3 cm diameter or greater with a prevailing pathology (e.g., as opposed to adenomyosis) of fibroids determined through ultrasound;
* Willing to maintain use or non-use of hormonal contraception from 3 months pre-study throughout the 12-month follow-up period;
* Willing to maintain use or non-use of anti-fibrinolytic agents from 3 months pre-study throughout the 12-month follow-up period;
* Able to tolerate the required prolonged supine position during treatment (approximately 6 hours);
* Willing and able to provide informed consent and to follow study-related requirements;

Exclusion Criteria:

* Pregnancy (as confirmed immediately prior to procedure)
* Fibroid diameter greater than 8.0 cm determined through transvaginal ultrasound; [or if 2 dimensions are measured, total dimension greater than 16 cm; or if the 3 dimensions (length, height, width) are measured, total dimension greater than 24 cm];
* Presence of a pedunculated fibroid determined by ultrasound; hysteroscopy, or saline infused sonography;
* Hydronephrosis as determined by radiologist interpretation on renal ultrasound pre-procedurally;
* Menopausal;
* Clinical history of any thromboembolic disease;
* Blood urine nitrogen (BUN) greater than 20 mg/dL and/or serum creatinine greater than 1.2 mg/dL unresolved with change in diet or hydration; · One or more lower uterine segment fibroids determined through pelvic exam;
* History of gynecologic malignancy, atypical endometrial hyperplasia, or pelvic inflammatory disease;
* Abnormal endometrial biopsy within the last 6 months prior to procedure;
* Pelvic mass outside the uterus suggesting other disease processes;
* Any current acute or chronic systemic infection or localized pelvic infection, including an unresolved urinary tract infection;
* Using GnRH agonist or mifepristone within 6-months prior to the start of the study;
* An intrauterine device (IUD) in place;
* Using anticoagulation therapy (except OTC treatments (e.g. aspirin)), or have an underlying bleeding disorder;
* Unsuitable for MRI examination, if within study subgroup to undergo MRI evaluation (e.g. severe claustrophobia, non-MRI-compatible implanted metalloid devices);
* Prior endometrial ablation, uterine artery embolization, or uterine artery ligation;
* Poor procedural candidate due to medical conditions as determined by the investigator (e.g. anesthesia class, renal insufficiency, heart disease);
* Grade 1 for 3D Color Doppler or no flow observed for cystoscopy on ureter flow assessment if applicable.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piet Hinoul, M.D., Study Director — Ethicon, Inc.
Locations (11):
- United States (9):
  - Women's Health Research, Phoenix, Arizona
  - Holy Cross Medical Group, Fort Lauderdale, Florida
  - University Women's Care - Wayne State University, Southfield, Michigan
  - Minnesota Gynecology and Surgery, Edina, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - North Carolina Children's & Adults' Clinical Research Foundation, Chapel Hill, North Carolina
  - Complete Healthcare for Women, Columbus, Ohio
  - Hahnemann University Hospital - Drexel University School of Med., Philadelphia, Pennsylvania
  - Matlock Ob/Gyn, Arlington, Texas
- St. Joseph's Health Care, London, Ontario, Canada
- Hospital Universitario, Monterrey, Nuevo León, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from June 2007 through May 2009. Sites included hospitals, surgical centers and private practices in North America.
Period: Overall Study
Arm/Group | DUAO Device
Started | 87
Completed | 60
Not Completed | 27
Not completed — Lost to Follow-up | 9
Not completed — Surgical re-intervention | 7
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | DUAO Device
Number analyzed (Participants) | 87
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 48
  Mexico | 30
  Canada | 9

OUTCOME MEASURES:

1. Primary Outcome: No Surgical Re-intervention
Description: Number of participants without any subsequent surgical procedure intended to manage fibroid symptoms performed. Potential procedures included surgical hysterectomy or dilatation and curettage (D&C) for treatment of menorrhagia; uterine artery embolization (UAE) or laparoscopic uterine artery occlusion; endometrial resection or ablation; myomectomy or myolysis.
Time Frame: Study completion
Population: ITT (Data missing for 5 participants)
Measure: Number; unit: participants
Groups:
- DUAO Device: Doppler-guided uterine artery occlusion device
Arm/Group | DUAO Device
Number analyzed (Participants) | 82
participants | 74 [82.7 to 95.9]

2. Primary Outcome: Improvement in Pictorial Blood Loss Assessment Chart (PBLAC) Score
Description: Number of participants with a 50% or greater reduction in PBLAC score from baseline at 12 mo and a PBLAC score of less than 250. PBLAC is a simple validated semiquantitative method of measuring total menstrual blood loss using a pictorial representation of blood loss, where higher scores indicate more blood loss. This hybrid endpoint combined the reduction in PBLAC score with the total PBLAC score.
Time Frame: From baseline to 12 months
Population: ITT (No data for 18 participants)
Measure: Number; unit: participants
Arm/Group | DUAO Device
Number analyzed (Participants) | 69
participants | 15 [12.7 to 33.3]

3. Secondary Outcome: Mean Improvement in Health Related Quality of Life (HRQOL) Scores
Description: Participants categorized as "better" in the total UFS-QOL questionnaire, indicating an overall improvement in health-related quality of life. On this scale, higher scores are indicative of better quality of life, with a maximum(best)score of 100 and a minimum (worst)score of 0. "Better" was defined as a change of +12 or more from baseline at 12 mo.
Time Frame: From baseline to 12 months
Population: ITT (No data for 20 participants)
Measure: Number; unit: participants
Arm/Group | DUAO Device
Number analyzed (Participants) | 67
participants | 54

4. Secondary Outcome: Maintenance of Menses
Description: Number of participants with continuation of menstrual cycles without interruption for three consecutive months
Time Frame: 12 months
Population: ITT (No data for 30 participants)
Measure: Number; unit: participants
Arm/Group | DUAO Device
Number analyzed (Participants) | 57
participants | 53

5. Secondary Outcome: Procedural Satisfaction
Description: Number of participants with responses of either "satisfied" or "very satisfied" on a qualitative survey that ranged from "very dissatisfied" (worst) to "very satisfied" (best)
Time Frame: 12 months
Population: ITT (No data for 19 participants)
Measure: Number; unit: participants
Arm/Group | DUAO Device
Number analyzed (Participants) | 68
participants
  Undecided | 11
  Very Dissatisfied | 2
  Dissatisfied | 5
  Satisfied | 21
  Very Satisfied | 29

6. Secondary Outcome: Decrease in Fibroid Bulk
Description: Number of participants with a minimum 15% decrease in fibroid bulk based on independent magnetic resonance imaging (MRI) review from baseline at 12 mo.
  Note: As per protocol, MRIs were planned only for subjects 1 - 40, 81 - 120, and 161-200.
Time Frame: From baseline to 12-months
Population: ITT (Due to early termination, only 39 subjects had MRIs. No data for 8 participants.)
Measure: Number; unit: participants
Arm/Group | DUAO Device
Number analyzed (Participants) | 31
participants | 10

7. Secondary Outcome: Mean Improvement in Uterine Fibroid Symptom Quality of Life (UFS-QOL) Symptom Severity Scores
Description: Number of participants categorized as "better" in the UFS-QOL sympton severity questionnaire, indicating an overall improvement in fibroid related symptoms. On this scale, higher scores are indicative of increasing symptom distress, with a maximum(worst)score of 100 and a minimum (best)score of 0. "Better" was defined as a change of -11 or less from baseline at 12 mo.
Time Frame: From baseline to 12 months
Population: ITT (No data for 18 participants.)
Measure: Number; unit: participants
Arm/Group | DUAO Device
Number analyzed (Participants) | 69
participants | 55

ADVERSE EVENTS:
Time Frame: 3 years
Description: Due to early study termination the longest timeframe of a patient's study participation was 2 years and 9 days. The shortest timeframe of study participation was 11 months 9 days.
Arm/Group | DUAO Device
Serious Adverse Events (participants affected / at risk) | 4/87
Other Adverse Events (participants affected / at risk) | 37/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DUAO Device (N=87)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Medication Error (Injury, poisoning and procedural complications) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DUAO Device (N=87)
Nausea (Gastrointestinal disorders) | 10 (10)
Procedural pain (Injury, poisoning and procedural complications) | 5 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Headache (Nervous system disorders) | 7 (7)
Hydronephrosis (Renal and urinary disorders) | 9 (9)
Dysmenorrhea (Reproductive system and breast disorders) | 6 (7)
Vaginal Discharge (Reproductive system and breast disorders) | 9 (10)
Pelvic pain (Injury, poisoning and procedural complications) | 10 (13)

LIMITATIONS AND CAVEATS:
Study was terminated early because 6 mo interim analysis of parallel European study showed that device was not meeting the primary endpoint. Target enrollment was 200 subjects, but results are based on 87 subjects who were treated with the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less